CLINICAL TRIAL: NCT06738472
Title: Efficacy of Home-Based Posture Exercises as an Addition to Pharmacological Treatment in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Researcher, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AEU-FTR1
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; home-based therapy; pain; quality of life
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetin+home based therapy (Experimental): Participants in this arm will receive standard pharmacological treatment for fibromyalgia as prescribed by a physician, in addition to a structured home exercise program. The home exercise program will include stretching and strengthening exercises targeting the spinal and trunk muscles and will be performed according to the study protocol. Clinical outcomes and spinal posture and mobility will be assessed using the Spinal Mouse® device in upright standing, maximum trunk flexion, and maximum trunk extension positions at baseline and follow-up.
  Interventions: Other: home based exercises
- Duloxetin only (No Intervention): Participants in this arm will receive standard pharmacological treatment for fibromyalgia as prescribed by a physician, without any additional exercise intervention. Clinical outcomes and spinal posture and mobility will be assessed using the Spinal Mouse® device in upright standing, maximum trunk flexion, and maximum trunk extension positions at baseline and follow-up.

INTERVENTIONS:
Other: home based exercises — given exercises to the participants
  Arms: Duloxetin+home based therapy

SUMMARY:
This interventional study aimed to evaluate the effects of home exercise in addition to pharmacological treatment on pain threshold and spinal mobility in fibromyalgia patients.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic pain syndrome characterized by widespread musculoskeletal pain, altered pain processing, fatigue, and functional limitations. In addition to pain-related symptoms, individuals with FM frequently present with postural alterations, reduced spinal mobility, and impaired segmental control of the spine, which may contribute to functional disability and reduced quality of life. However, objective assessment of spinal posture and segmental mobility in FM remains limited.

This study aims to comprehensively evaluate spinal posture and sagittal plane mobility in patients with fibromyalgia using the Spinal Mouse®, a validated, non-invasive, computer-assisted device that measures spinal curvature and segmental inclination without radiation exposure. The Spinal Mouse allows for reliable assessment of thoracic and lumbar spinal alignment as well as dynamic movement patterns during functional tasks.

ELIGIBILITY:
Inclusion Criteria:

* Participants were between the ages of 18 and 65,
* No diagnosis of rheumatic disease,
* No diagnosis of chronic comorbid disease,
* Participants diagnosed with fibromyalgia syndrome according to the European League Against Rheumatism (EULAR) criteria will be included as volunteers.

Exclusion Criteria:

* Patients under 18, over 65 years of age
* Those diagnosed with chronic comorbid diseases
* Those with a history of rheumatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-28 (Actual)

PRIMARY OUTCOMES:
Algometry | 4 weeks
  pain pressure threshold
Spinal mouse for spinal mobility | 4 weeks
  spinal range of motion

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 4 weeks
  used to assess anxiety and depressive symptoms in clinical populations
Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  Quality of Sleep
Short form-12 (SF-12) | 4 weeks
  Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozcelep OF, Ustun I, Algun ZC. Effect of task-oriented training on pain, functionality, and quality of life in rheumatoid arthritis. Turk J Phys Med Rehabil. 2022 Mar 1;68(1):76-83. doi: 10.5606/tftrd.2022.6666. eCollection 2022 Mar. PMID 35949976